CLINICAL TRIAL: NCT07058649
Title: Individualized Downstaging Prediction Model for HCC Beyond the UCSF Criteria
Brief Title: Downstaging Prediction Model for HCC
Status: Not yet recruiting | Type: Observational
Sponsor: Beijing Tsinghua Chang Gung Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 25288-0-02
Record Dates: First submitted 2025-07-01; First posted 2025-07-10 (Actual); Last update posted 2025-07-10 (Actual); Status verified 2025-07

CONDITIONS: HCC - Hepatocellular Carcinoma
Keywords: downstaging; UCSF
MeSH Terms: conditions — Carcinoma, Hepatocellular

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Successful downstaging: Failure downstaging

SUMMARY:
This study is a real-world, single-center study that collects imaging and clinical data from patients with HCC who are downstaged beyond the UCSF criteria.

DETAILED DESCRIPTION:
This study is a real-world, single-center study that collects imaging and clinical data from patients with HCC who are downstaged beyond the UCSF criteria. It constructs a predictive model for downstaging treatment of liver cancer beyond the UCSF standards and completes external validation. This model will assist in clinical decision-making for the downstaging treatment of liver cancer beyond the UCSF criteria. Further downstaging methods are stratified to guide the selection of individualized downstaging treatment options for liver cancer beyond the UCSF standards.

ELIGIBILITY:
Inclusion Criteria:

* (A) Adult patients with HCC over the age of 18 (clinically diagnosed or pathologically diagnosed); (B) Liver function Child-Pugh score of Class A, or Class B with a score of 7 or below (including 7); (C) A single solid tumor with a diameter of ≥6.5 cm; three or more lesions, among which at least one tumor has a diameter >4.5 cm or the sum of the diameters is ≥8 cm; invasion of major blood vessels regardless of tumor size and number.

Exclusion Criteria:

* (A) Presence of distant metastasis outside the liver; (B) General performance status score (PS score) greater than 2 points.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: HCC patients beyond UCSF criteria
Sampling Method: Non-Probability Sample
Enrollment: 369 (Estimated)
Dates: Start 2025-07-16 (Estimated); Primary Completion 2027-10-01 (Estimated); Study Completion 2027-12-01 (Estimated)

PRIMARY OUTCOMES:
Downstagingoutcomes | 3 months after downstaging
  Successful downstaging is defined by meeting the UCSF criteria after downstaging; no invasion of the main trunk of the portal vein or the main trunk of the hepatic vein; and no lymph node invasion. The evaluation criteria used for interpretation are the mRECIST (modified Response Evaluation Criteria in Solid Tumors) standards.

IPD SHARING:
Plan to Share IPD: Undecided